CLINICAL TRIAL: NCT01889199
Title: Androgen Excess as a Cause for Adipogenic Dysfunction in PCOS Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Daniel A. Dumesic, MD, Professor, Division of Reproductive Endocrinology and Infertility, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UCLA IRB #12-001780
Record Dates: First submitted 2013-06-20; First posted 2013-06-28 (Estimated); Results first posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-12

CONDITIONS: Polycystic Ovary Syndrome (PCOS)
Keywords: polycystic ovary syndrome; hirsutism; anovulation; oligomenorrhea; amenorrhea; hyperandrogenism; antiandrogen effect
MeSH Terms: conditions — Polycystic Ovary Syndrome; Hirsutism; Anovulation; Oligomenorrhea; Amenorrhea; Hyperandrogenism | interventions — Flutamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sugar pill (Placebo Comparator): Placebo intervention
  Interventions: Other: Placebo
- Flutamide (Experimental): Flutamide 125 mg orally daily for six 28-day cycles.
  Interventions: Drug: Flutamide

INTERVENTIONS:
Drug: Flutamide — Flutamide 125 mg orally each 28 day cycle for 6 cycles
  Other Names: Euflex
  Arms: Flutamide
Other: Placebo — Placebo orally each 28 day cycle for 6 cycles
  Arms: Sugar pill

SUMMARY:
The purpose of this research study is to collect specimen samples and study medical information from women with Polycystic Ovary Syndrome (PCOS) and women without PCOS. The goal is to learn more about the changes that take place in the body that result in PCOS.

We anticipate that 32 women will take part in this study (16 without PCOS and 16 with PCOS). All patients will undergo a physical exam, blood tests, and ultrasound of their ovaries. If they meet the criteria for this study, they will then undergo additional blood tests, removal of a small amount of subcutaneous abdominal fat, measurement of regional body fat (i.e., DXA scan) and a modified frequently-sampled intravenous glucose tolerance test (FSIGTT). The women without PCOS will complete the study at this point.

The women with PCOS will be randomized to receive the drug flutamide 125 mg/day or placebo. They will take the drug every day for six 28-day cycles. They will be asked to collect and store a urine sample once a week. They will also be asked to complete a pill diary and menstrual diary. Once a month while they are taking the flutamide/placebo, they will return to the clinic and bring their frozen urine samples. At that time they will undergo a physical exam, toxicity assessment, and blood draw.

Quality of Life assessments will be done at the beginning of the study for all participants. Women with PCOS who are taking the flutamide or placebo will be asked to repeat the Quality of Life assessments during the study and at the end of the study.

After the six 28-day cycles are completed they will then undergo additional blood tests, removal of a small amount of subcutaneous abdominal fat, measurement of regional body fat (i.e., DXA scan) and a modified frequently-sampled intravenous glucose tolerance test (FSIGTT).

Six months following the completion of all study protocol procedures, participants who received flutamide/placebo will be contacted by phone to check on the status of their health. They will be asked if they have experienced any health problems or have become pregnant since they completed the study procedures.

DETAILED DESCRIPTION:
Aim 1. Examine mechanisms of subcutaneous abdominal adipose (fat) development in normal-weight PCOS women vs. BMI- and age-matched normal (control) women.

Subjects and clinical assessment: We will recruit 16 lean (18.5-25 kg/M2) PCOS subjects and 16 age- and BMI-matched controls. Subjects will complete a standardized questionnaire emphasizing menstrual dating, abnormal hair growth and acne. The questionnaire also will annotate age, smoking status, medications, surgical history and family histories of excess hair growth in female relatives and of diabetes in parents or siblings for exclusion criteria and for inclusion of some basic traits as covariates. Subjects also will undergo a physical examination; hirsutism will be scored by the modified Ferriman-Gallwey (mFG) method. Transvaginal sonography (TVUS) will be performed to determine the presence or absence of polycystic ovaries. A screening blood sample will be obtained for determinations of steroid hormones, SHBG, TSH, and prolactin.

Women of any ethnicity between the ages of 18 and 35 years will be recruited. PCOS patients will be diagnosed by 1990 NIH criteria. Controls will have regular menstrual cycles at 21 to 35 day intervals, a luteal phase progesterone (P4) level > 3 ng/mL, and no evidence of hirsutism, acne, alopecia, polycystic ovaries or endocrine dysfunction. Exclusion criteria are: present/past history (<1 year) of smoking, cancer, alcohol abuse, drug addiction, severe depression, or post traumatic stress; diabetes; uncontrolled hypertension (≥ 165/100); clinically significant hepatic or renal disease, or other major medical illness; signs or symptoms of infection; recent (within 30 days) use of an experimental device; recent (within 3 months) use of androgens, anabolic steroids or non-steroidal anti-inflammatory drugs; recent (within 3 months) use of hormonal agents (including birth control pills or insulin sensitizers); use of the drug warfarin.

Studies will be conducted in the follicular phase in controls and during amenorrhea in PCOS women. All subjects will undergo a modified frequently-sampled intravenous glucose tolerance test (FSIGTT). Glucose in the form of a 50% solution (0.3 g/kg) and regular human insulin (0.03 units/kg) will be injected through an intravenous line at 0 and 20 min, respectively. Blood will be collected at -20, -15, -5, 0, 2, 4, 8, 19, 22, 30, 40, 50, 70, 90, and 180 min for glucose and insulin determinations. Mathematical modeling of serial glucose and insulin determinations will calculate: insulin sensitivity index (SI, i.e. the action of insulin to accelerate glucose uptake and suppress glucose production), glucose effectiveness index (SG, i.e. the combined effect of glucose to enhance glucose uptake and suppress endogenous glucose production at basal insulin levels) and the acute response to glucose (AIRG).

Adipocytes isolation and culture: Approximately 1-2 gms of fat will be obtained from the lower SC abdomen using standard procedures under local anesthesia. Adipocytes (fat cells) and surrounding fat tissue will be isolated to measure adipocyte cell number and diameter, lipid accumulation and function, adiponectin, and stem cell development.

Procedures: All procedures will be performed in normal and PCOS women at the start of study.

i). Venipuncture: Fasting blood will be collected for blood count, chemistry panel, LH, FSH, total/free T, DHT, A4, DHEAS, E1, E2, anti-mullerian hormone (AMH), SHBG, adiponectin, leptin, IL-6, lipid profile and free fatty acids (FFAs).

ii ). Body composition: Body composition will be assessed by BMI, waist-to-hip circumference and DEXA scanning. Girths will be measured at the waist (narrowest section of the torso between ribs and umbilicus) and hips (largest protrusion of the hip region, above the gluteal fold). For total body fat and regional fat distribution, whole body scans will be performed, utilizing DEXA imaging.

iii). Body fat distribution: Total body DEXA will measure abdominal fat (i.e., the area between the dome of the diaphragm and the top of the hip. Total body DEXA images also will determine % body fat; fat-free body mass; total body, abdominal, and leg fat; and abdomen/leg fat mass ratio. The leg region is that area below the top of the hip bone (greater trochanter).

iv). Ovarian testing: Transvaginal ultrasound will be performed in the follicular phase in controls and during amenorrhea in PCOS women. Ovarian volume will be calculated. Antral follicle number, defined as the total follicle number (2-9 mm in diameter) of both ovaries, will be determined by 1 investigator (D.A.D.). Polycystic ovaries will be identified, with one such ovary sufficient to define PCO

Aim 2. Determine the role of androgen in SC abdominal ASC dysfunction and its relation to metabolism in normal-weight PCOS women through androgen. antagonism by clinical use of flutamide vs. placebo.

Modified FSIGTT and Adipogenic studies: The modified FSIGTT and all adipogenic studies performed at study initiation will be repeated at the end of the 6-month flutamide vs. placebo intervention in PCOS women.

Procedures: All procedures performed at study initiation also will be repeated at the end of the six 28-day cycles of flutamide vs. placebo intervention in PCOS women. In addition, monthly liver function studies will be performed to detect possible elevations of serum transaminase levels above the normal range during flutamide vs. placebo therapy.

Menstrual records: Ovulatory frequency will be determined by having subjects keep a daily menstrual record and collect weekly first morning urine samples for possible progesterone and creatinine determinations. Urine samples will be frozen for later analysis to determine evidence of ovulation, as necessary.

Aim 3. Identify epigenetic changes that underlie SC abdominal ASC dysfunction in normal-weight PCOS women vs. BMI- and age-matched controls.

Subcutaneous abdominal adipose stem cells from PCOS and control women will be grown into newly-formed fat cells (adipocytes) in the laboratory. Cells will be studied before and after 6-month treatment with placebo vs flutamide for changes in the cell epigenome (methylation, RNA sequences and histone modification).

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18 to 35 years.

Groups will be: 16 lean controls and 16 age- and BMI-matched PCOS women randomized to flutamide vs. placebo for 6 months.

i) Lean patients with PCOS: 16 subjects with PCOS (defined by 1990 NIH criteria [all Aims]), BMI 18.5-25 kg/m2. This BMI range is defined as normal and has been chosen to examine underlying mechanisms of PCOS-related androgen excess in the genesis of adipogenic and ovarian dysfunction, independent of obesity.

ii) Lean control women: 16 healthy subjects, BMI 18.5-25 kg/m2. Controls will have regular menstrual cycles, and no evidence of hirsutism, acne, alopecia, polycystic ovaries, and/or endocrine dysfunction. This BMI range has been chosen to match that of the PCOS group.

Exclusion Criteria:

* Exclusion criteria for study participation are: present or past history (<1 years) of smoking, cancer, alcohol abuse, drug addiction, severe depression, or post traumatic stress; diabetes; uncontrolled hypertension (≥ 165/100); clinically significant hepatic or renal disease, or other major medical illness; recent (within 3 months) use of androgens, anabolic steroids or hormonal agents (including birth control pills or insulin sensitizers). These exclusion criteria are chosen to avoid effects from medical conditions, environmental factors or exogenous agents. Women taking the drug warfarin, CYP active medications, or herbs will be excluded.

The screener will assess the participants response to establish if depression or drug use exclude participation in this study.

Women taking beta blockers will be excluded.

Women who have taken birth control pills or had a Mirena IUD or used Plan B contraception during the previous 3 months will be excluded.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2013-04; Primary Completion 2023-07-06 (Actual); Study Completion 2023-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Dumesic, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCaliforniaLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dumesic DA, Winnett C, Lu G, Grogan TR, Abbott DH, Naik R, Chazenbalk GD. Randomized clinical trial: effect of low-dose flutamide on abdominal adipogenic function in normal-weight women with polycystic ovary syndrome. Fertil Steril. 2023 Jan;119(1):116-126. doi: 10.1016/j.fertnstert.2022.09.324. Epub 2022 Nov 15. PMID 36400597

RESULTS

PARTICIPANT FLOW:
Groups:
- Age- and Body Mass Index-matched Controls: Baseline measures assessed on non-PCOS controls
Period: Overall Study
Arm/Group | Sugar Pill | Flutamide | Age- and Body Mass Index-matched Controls
Started | 6 | 5 | 12
Baseline | 6 | 5 | 12
6-month Assessment on Intervention Arms | 6 | 5 | 0
Completed | 6 | 5 | 0
Not Completed | 0 | 0 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar Pill | Flutamide | Age- and Body Mass Index-matched Controls | Total
Number analyzed (Participants) | 6 | 5 | 12 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 12 | 23
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 12 | 23
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 4 | 4 | 14
  Unknown or Not Reported | 0 | 1 | 8 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 6 | 4 | 3 | 13
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 8 | 8
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Lipid Content of PCOS Subcutaneous (SC) Abdominal Adipocytes Matured in Vitro.
Description: Lipid content of PCOS subcutaneous (SC) abdominal stem cells during adipocyte maturation in vitro at baseline and after 6 months treatment
  Lipid staining and immunofluorescence:
  Newly-formed adipocytes were fixed and stained with Oil-Red-O (Sigma Aldrich, St. Louis, MO) for 20 min at room temperature to visualize lipid droplets. Nuclei were identified by the nuclear staining marker 4',6-diamidino-2-phenoylidole (DAPI) (1:3000 [Invitrogen, Carlsbad, CA]). After 4 washes with deionized water, lipid staining was quantified by immunofluorescence. Twenty representative images were taken of fluorescent cells with an EVOS FL Digital Inverted Fluorescence microscope (Westover Scientific Inc, Bothell, WA) and fluorescence units/cell number were quantified using ImageJ software (NIH, Bethesda, MD).
Time Frame: Baseline, 6 months
Population: Assessed for participants with PCOS
Measure: Mean (Standard Deviation); unit: fluorescence units/cell number
Arm/Group | Sugar Pill | Flutamide | Age- and Body Mass Index-matched Controls
Number analyzed (Participants) | 6 | 5 | 0
fluorescence units/cell number
  Baseline | 2.0 (0.6) | 5.6 (4.1) |
  6 months | 1.37 (0.7) | 3.8 (3.9) |
  Change | -0.6 (0.4) | -1.8 (0.6) |
Statistical Analysis 1: Comparison: Sugar Pill vs Flutamide; Only PCOS women were randomized to flutamide versus placebo; controls were not randomized A sample size of 11 per group (PCOS women versus controls) provided adequate power (approximately 80%) to detect effect sizes as small as 1.25 using a two-sample t-test (alpha=0.05, 2 tailed). A sample size of 5 per group (flutamide-treated versus placebo-treated PCOS women) also gave adequate power (approximately 80%) to detect effect sizes as small as 2 using a two-sample t-test (alpha=0.05, 2 tailed); Test type: Other; p = 0.004, t-test, 2 sided — a priori threshold p<0.05; Mean Difference (Final Values) = 1.12

2. Secondary Outcome: Fasting Glucose Levels
Description: Fasting glucose levels at baseline for all participants, and at 6 months for intervention arms
Time Frame: Baseline, 6 months
Population: Control group was assessed at baseline only
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Sugar Pill | Flutamide | Age- and Body Mass Index-matched Controls
Number analyzed (Participants) | 6 | 5 | 12
mg/dL
  Baseline | 85.6 (4.6) | 83.9 (4.8) | 85.8 (6.1)
  6 months: number analyzed (Participants) | 6 | 5 | 0
  6 months | 85.3 (4.8) | 88.6 (5.6) |
  Change: number analyzed (Participants) | 6 | 5 | 0
  Change | -0.3 (3.9) | 4.6 (1.6) |
Statistical Analysis 1: Comparison: Sugar Pill vs Flutamide; 6-month changes from baseline were compared between placebo- and flutamide-treated PCOS women using an unpaired Student's t-test to determine whether one group changed more than the other over this time interval; Test type: Other; Mean Difference (Net) = 0.024

3. Secondary Outcome: Depression as Assessed by Beck Depression Inventory (BDI)
Description: Number of participants with risk of severe depression as determined by 21 questions on a 4-point Likert scale, scores could range from 0-63, with higher score indicating a worse outcome. Scores above 30 indicate Severe depression, and scores above 40 indicate Extreme Depression.
Time Frame: 6 months
Population: Assessed only for intervention arms of healthy normal-weight PCOS women by NIH criteria
Measure: Count of Participants; unit: Participants
Arm/Group | Sugar Pill | Flutamide
Number analyzed (Participants) | 6 | 5
Participants | 0 | 0

4. Secondary Outcome: Percent Android Fat Mass
Description: Percent of abdominal (android) fat by Total body dual-energy x-ray absorptiometry (DXA) scan
Time Frame: Baseline, 6 months (intervention arms only)
Population: Control group was assessed at baseline only
Measure: Mean (Standard Deviation); unit: percent abdominal (android) fat mass
Arm/Group | Sugar Pill | Flutamide | Age- and Body Mass Index-matched Controls
Number analyzed (Participants) | 6 | 5 | 12
percent abdominal (android) fat mass
  Baseline | 6.0 (1.4) | 6.1 (1.8) | 5.5 (0.5)
  6 months: number analyzed (Participants) | 6 | 5 | 0
  6 months | 6.4 (1.2) | 5.9 (1.4) |
  Change: number analyzed (Participants) | 6 | 5 | 0
  Change | 0.4 (0.4) | -0.3 (0.5) |
Statistical Analysis 1: Comparison: Sugar Pill vs Flutamide; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.040, t-test, 2 sided; Mean Difference (Net) = 0.040

5. Secondary Outcome: Fasting Serum Lipoprotein Levels
Description: Fasting serum low-density lipoprotein levels at baseline and (for intervention arms only) after 6 months
Time Frame: 6 months
Population: Control group was assessed at baseline only
Measure: Mean (Standard Deviation); unit: (log)mg/dL
Arm/Group | Sugar Pill | Flutamide | Age- and Body Mass Index-matched Controls
Number analyzed (Participants) | 6 | 5 | 12
(log)mg/dL
  Log triglyceride - Baseline | 1.9 (0.3) | 1.7 (0.1) | 1.7 (0.1)
  Log triglyceride - 6 months: number analyzed (Participants) | 6 | 5 | 0
  Log triglyceride - 6 months | 1.9 (0.4) | 1.7 (0.2) |
  Log triglyceride - Change: number analyzed (Participants) | 6 | 5 | 0
  Log triglyceride - Change | 0.0 (0.1) | 0.0 (0.1) |
  Log non-high-density lipoprotein baseline | 2.0 (0.1) | 2.0 (0.1) | 1.94 (0.10)
  Log non-high-density lipoprotein - 6 months: number analyzed (Participants) | 6 | 5 | 0
  Log non-high-density lipoprotein - 6 months | 2.0 (0.1) | 2.0 (0.1) |
  Log non-high-density lipoprotein - change: number analyzed (Participants) | 6 | 5 | 0
  Log non-high-density lipoprotein - change | 0.0 (0.0) | -0.1 (0.1) |
  Log low-density lipoprotein - Baseline | 1.8 (0.1) | 2.0 (0.1) | 1.88 (0.10)
  Log low-density lipoprotein - 6 months: number analyzed (Participants) | 6 | 5 | 0
  Log low-density lipoprotein - 6 months | 1.8 (0.1) | 1.9 (0.1) |
  Log low-density lipoprotein - Change: number analyzed (Participants) | 6 | 5 | 0
  Log low-density lipoprotein - Change | 0.0 (0.0) | -0.1 (0.1) |
Statistical Analysis 1: Comparison: Sugar Pill vs Flutamide; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.034, t-test, 2 sided

6. Other Pre Specified Outcome: Number of Participants Experiencing Elevated Liver Transaminases (Serum Glutamic Oxaloacetic Transaminase [SGOT]; Serum Glutamic-pyruvic Transaminase [SGPT])
Description: This study carefully considers the safety of low-dose flutamide in examining how hyperandrogenism in PCOS affects ovarian function, subcutaneous fat storage and glucose metabolism. The 125 mg oral dose of flutamide has been specifically chosen because it has not been associated with liver enzyme abnormalities (0%, 62.5-125 mg/day), while being as effective as high dose flutamide in improving androgenic symptoms. Furthermore, in the rare event mild elevation of hepatic enzymes occurs with low-dose flutamide despite its dose-dependency, it is easily detected and reversible.
Time Frame: 6 months
Population: Assessed only for intervention arms of healthy normal-weight PCOS women by NIH criteria
Measure: Count of Participants; unit: Participants
Arm/Group | Sugar Pill | Flutamide
Number analyzed (Participants) | 6 | 5
Participants | 0 | 0

7. Secondary Outcome: Fasting Serum Total Cholesterol
Description: Fasting serum total cholesterol at baseline and (for intervention arms only) after 6 months
Time Frame: Baseline, 6 months
Population: Control group was assessed at baseline only
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Sugar Pill | Flutamide | Age- and Body Mass Index-matched Controls
Number analyzed (Participants) | 6 | 5 | 12
mg/dL
  Total cholesterol - Baseline | 153.7 (29.1) | 184.0 (27.0) | 153.0 (21.7)
  Total cholesterol - 6 months: number analyzed (Participants) | 6 | 5 | 0
  Total cholesterol - 6 months | 155.3 (31.6) | 168.0 (14.7) |
  Total cholesterol - Change: number analyzed (Participants) | 6 | 5 | 0
  Total cholesterol - Change | 1.7 (9.4) | -16.0 (24.4) |

ADVERSE EVENTS:
Time Frame: Baseline-6 months (intervention arms only), Baseline-only collection for control arm
Arm/Group | Sugar Pill | Flutamide | Age- and Body Mass Index-matched Controls
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5 | 0/12
Other Adverse Events (participants affected / at risk) | 0/6 | 0/5 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-07): https://cdn.clinicaltrials.gov/large-docs/99/NCT01889199/Prot_SAP_000.pdf
  • Informed Consent Form (2020-02-26): https://cdn.clinicaltrials.gov/large-docs/99/NCT01889199/ICF_001.pdf